CLINICAL TRIAL: NCT05298930
Title: A Feasibility Study Evaluating Connected Bikes as a Means of Adapted Physical Activity in Children, Adolescents and Young Adults Requiring Hematopoietic Stem Cell Transplantation
Brief Title: Feasibility Study to Assess an Adapted Physical Activity Program in Children, Adolescents and Young Adults Requiring Hematopoietic Stem Cell Transplantation
Acronym: EVAADE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: EVAADE ET 21-015
Record Dates: First submitted 2022-03-03; First posted 2022-03-28 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2023-08

CONDITIONS: Haematological Malignancy; Acute Leukemia; Myelodysplastic Syndromes; Hemoglobinopathy in Children; Bone Marrow Aplasia; Severe Combined Immunodeficiency
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Anemia, Aplastic; Severe Combined Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical activity intervention (Experimental): The intervention will take place during the whole isolation phase and will consist of an APA program defined at inclusion, integrating supervised sessions with an APA teacher, as well as unsupervised sessions. The program will be individualized according to the patient's age, physical condition and PA preferences. The sessions will also be adapted to the biological, psychological and social parameters of the patients.
  The intervention will be carried out during the entire hospitalization period and for a maximum of 3 months. An connected bike will be installed in the patient's room for the duration of the hospitalization.
  Interventions: Other: Physical activity program

INTERVENTIONS:
Other: Physical activity program — The supervised sessions will be offered 4 times a week in the participants' rooms by the APA teachers and will include moderate intensity aerobic activities (exercise bike), muscle strengthening (dumbbells, elastic bands, medicine balls) and playful situations (ball games, cooperative games, body expression games).
  Each patient will also be able to perform unsupervised sessions (on their own), following the advice given by the APA teacher. These unsupervised sessions can be done independently on the bike.
  In order to encourage patients to perform these unsupervised sessions, patients and their relatives will be given a connected device and will have access to a mobile application developed by the Kiplin company, which offers connected physical activity games to be performed in teams (from 2 to 4 participants). These games, lasting from 1 to 3 weeks, use the participants' daily PA level as a unit of animation and are punctuated by challenges.

SUMMARY:
Allogeneic haematopoietic stem cell transplantation (aHSCT) is the only curative treatment for many paediatric and young adult haematological pathologies (acute leukaemia, myelodysplastic syndromes haemoglobinopathies, bone narrow aplasia, severe combined immunodeficiency). Despite the major therapeutic progress made over the last 50 years, particularly in terms of supportive care, post-transplant morbidity and mortality remain high. Infectious complications, whose incidence varies between 30 and 60%, are the first cause of mortality in the immediate post-transplant period.

In order to protect the patient from the occurence of severe infectious episodes, aHSCT must be performed in a highly protected environment (positive pressure chambers).

This has consequences for the experience and impact of hospitalization on the patient and family. This is particularly true in pediatrics, with children, adolescents or young adults, where it is not only the patient's quality of life that is at stake, but also his emotional and psychomotor development. In this specific population, prolonged hospitalization (at least 6 weeks) in a sterile room will be responsible for physical deconditioning accompanied by a decrease in muscle mass. Patients often experience an deteriorated quality of life.

Today, the benefits of physical activity (PA) during and after cancer treatment have been widely demonstrated.

The objective of the study is to assess the feasibility of an adapted physical activity program during the isolation phase for achieving aHSCT in children, adolescents and young adults. This is a prospective, interventional, monocentric cohort study conducted at the institute of Paediatric Haematology and Oncology in Lyon. The intervention will take place during the isolation phase and will be based on an adapted physical activity (APA) program defined at inclusion, integrating supervised sessions with an APA teacher, as well as autonomous sessions performed by means of a connected bike in the sterile room. The program will be individualized according to age, aerobic capacities, and PA preferences. Sessions will also be tailored to the biological, psychological, and social parameters of patients.

The total duration of the intervention is 3 months. To date, no PA studies have been performed in patients under 21 years old requiring aHSCT during the sterile isolation phase. EVAADE will therefore be the first study in this population to offer an innovative procedure with a connected device.

ELIGIBILITY:
Inclusion Criteria:

* 8 years ≤ Age ≤ 21 years
* Height ≥ 110 cm
* Histologically or cytologically confirmed malignant or non-malignant haemopathy
* Indication for hematopoietic stem cell transplantation
* Hospitalization in a sterile room in the investigating center
* Certificate of no contraindicatication to practice an APA, issued by the oncologist or the attending physician
* Having a smartphone available in the sterile room (iOS version 12 (iPhone/Apple) or 6 under Android at least) for playing connected games
* Signed and dated written consent (patient or parents of minor patients with obtaining the minor's acceptance)

Exclusion Criteria:

* Severe heart disease and uncontrolled cardiovascular disease

Temporary contraindications

* Severe anemia (hemoglobin ≤ 8 g/dl) will need to be treated (transfusion of red blood cells [RBCs]) before resuming the physical activity program.
* Severe infectious syndrome in progress and/or febrile feeling with accompanying signs (productive cough, muscle pain).

Inclusion criteria for relatives :

* Person visiting the patient in a sterile room during the hospital stay
* At least 8 years old
* Height ≥ 110 cm
* Have a smartphone (iOS version 12 (iPhone/Apple) or 6 under Android at least) for the realization of the connected games.
* Not having any contraindication to physical activity.
* Signed and dated written consent (minor's relative or parents with the minor's acceptance).

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
observance to the physical activity program | 3 months
  achieved/non achieved (achieved meaning the patient attended at least one session of 15 minutes weekly during the whole program, considering both supervised and unsupervised sessions)

SECONDARY OUTCOMES:
Impact of unsupervised sessions on patients' PA practice | baseline, 3 months
  Rate of unsupervised sessions/total of performed sessions
Impact of the physical activity program on weight | baseline, 3 months
  weight in kgs
Impact of the physical activity on waist circumference | baseline, 3 months
  waist circumference assessed in cm
Impact of the physical activity program on hip circumference | baseline, 3 months
  hip circumference assessed in cm
Impact of the physical activity program on body mass index | baseline, 3 months
  weight/(size)^2
Impact of the physical activity program on endurance capacity | baseline, 3 months
  Harvard step test
Impact of the physical activity program on muscle strength | baseline, 3 months
  Dynanometer
Impact of the physical activity program on fatigue | baseline, 3 months
  Visual analogic scale from 0 to 10
Self efficacy feeling | 3 months
  HAPA questionnaire
Motivation towards physical activity | baseline, 3 months
  BREQ-2 questionnaire
Impact of the PA program on metabolic syndrome | baseline, 3 months
  Lipid check-up
Impact of social environment of PA practice | 3 months
  PA practice of patient / PA practice of relatives
Overall satisfaction | 3 months
  Likert-scale questionnaire
Acceptability of the intervention | baseline
  Number of enrolled patients/number of eligible patients

CONTACTS AND LOCATIONS:
Locations (1):
- Institut d'Hématologie et d'Oncologie Pédiatrique, Lyon, France

IPD SHARING:
Plan to Share IPD: No